CLINICAL TRIAL: NCT04415931
Title: Local Infiltration Analgesia Vs. Interscalene Block in Total Shoulder Arthorplasty: A Randomized Controlled Trial
Brief Title: Local Infiltration Analgesia Vs. Interscalene Block in Total Shoulder Arthorplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, H. Mike Kim, ASSOCIATE PROFESSOR OF CLINICAL ORTHOPAEDIC SURGERY, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022248
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Osteoarthritis; Cuff Tear Arthropathy; Massive Rotator Cuff Tear
Keywords: Total Shoulder arthroplasty; Reverse Shoulder arthroplasty; Cuff tear arthropathy; massive irreparable rotator cuff tear; Anatomic total shoulder arthroplasty; Shoulder osteoarthritis
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomized prior to their scheduled surgery date by our research team using a randomization protocol developed by our department biostatistics team. The surgeons and anesthesiologists will be blinded about the group assignment until the day before surgery. The group assignment will be sealed in an envelope and delivered to the surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local infiltration analgesia group (Experimental): This group of patients will receive local infiltration analgesia
  Interventions: Procedure: Local infiltration analgesia
- Interscalene block group (Active Comparator): This group of patients will receive interscalene block
  Interventions: Procedure: Interscalene block

INTERVENTIONS:
Procedure: Local infiltration analgesia — Local infiltration injection intraoperatively prior to closing during the procedure. A standardized dose of 100 mL of infiltration will be utilized according to the following formula. The mixture will be injected into the deltoid and pectoralis major muscles and fasciae, and subcutaneous tissues using an 18-guage needle.
  Total dose 100mL
  Ropivacaine 0.5% 40mL Epinephrine 1mg/mL 0.1mL Ketorolac 30mg/mL 1mL Morphine 10mg/mL 0.5mL Normal saline 0.9% 58.4mL
  Arms: Local infiltration analgesia group
Procedure: Interscalene block — Standard interscalene brachial plexus regional block
  Arms: Interscalene block group

SUMMARY:
Pain management following total shoulder arthroplasty is an important factor in determining patient outcomes and satisfaction. Interscalene brachial plexus blockade has been used successfully to minimize pain in the acute post-operative period. While shown to be effective, interscalene blockade has known complications. In addition, interscalene block has been shown to be significantly more expensive when compared to local anesthesia infiltration.

Local anesthetics such as bupivacaine have long been used to assist in post-operative anesthesia. Recent reports have demonstrated local infiltration of liposomal bupivacaine to be similar to interscalene block in regards to patient analgesia even in the first 24 hours post operatively, with the added benefit of lower complications and costs. While most reports examine the efficacy of local infiltration with liposomal bupivacaine in the shoulder, other total joint literature has been positive regarding the use of local infiltration analgesic mixture for improved post-operative analgesia using a multi-modal approach to infiltrative analgesia. Despite these reports, the role and efficacy of local infiltration analgesia in shoulder arthroplasty is lacking. The purpose of the proposed study is to determine the efficacy and safety of local infiltration analgesia in shoulder arthroplasty in comparison to interscalene block through a randomized prospective clinical trial. Our hypothesis is that local infiltration analgesia will lead to postoperative pain scores, opiate consumption, and complication rate that are not significantly different from interscalene block.

DETAILED DESCRIPTION:
1. SELECTION OF SUBJECTS • Inclusion Criteria: Adult patients (18 years of age or greater) undergoing primary anatomic or reverse total shoulder arthroplasty secondary to osteoarthritis, cuff tear arthropathy, or massive irreparable rotator cuff tear.

   • Exclusion Criteria :
   * Narcotic dependent
   * Previous ipsilateral open shoulder surgery
   * Chronic pain syndromes (fibromyalgia)
   * Contraindication to regional anesthesia
   * Cervical radiculopathy
   * Unable to give consent; Prisoner
   * Workers compensation insurance
   * Mentally Disabled.
   * Pregnant Patients
2. STUDY PROCEDURE • Timeline: 2 weeks of data collection

   • Study subjects: Study candidates will be identified as they present to the clinic at the Missouri Orthopaedic Institute at the University of Missouri, and will be evaluated by the principle investigator. Informed consent will be obtained as per IRB protocol. Enrollees will receive a copy of the study protocol, consent, and HIPAA form. Background patient information will be collected including age, sex, BMI and co-morbidities. American Society of Anesthesiologist (ASA) classification will be assigned by the involved anesthesiologist.

   Interscalene regional block is routinely administered at our institution prior to total shoulder arthroplasty. Patients will be randomized prior to their scheduled surgery date by our research team using a randomization protocol developed by our department biostatistics team. The surgeon and surgical assistants will be blinded about the group assignment until the morning of the surgery day. The group assignment will be sealed in an envelope and delivered to the surgeon. If randomized to the interscalene block group, the anesthesia team will administer the block preoperatively in routine fashion. The standard anesthesia protocol for total shoulder arthroplasty patients is as follows:

   • Preoperative: Acetaminophen 1000mg PO Gabapentin 300mg PO Interscalene block: 3-5mL of 0.5% bupivacaine plus 10mL Exparel (1-2 mg of midazolam and/or 50-100 mcg of fentanyl IV for sedation)

   If randomized to local infiltration analgesia, the patient will receive local infiltration injection intraoperatively prior to closing during the procedure. A standardized dose of 100 mL of infiltration will be utilized according to the following formula. The mixture will be injected into the deltoid and pectoralis major muscles and fasciae, and subcutaneous tissues using an 18-guage needle.

   Total dose 100mL Ropivacaine 0.5% 40mL Epinephrine 1mg/mL 0.1mL Ketorolac 30mg/mL 1mL Morphine 10mg/mL 0.5mL Normal saline 0.9% 58.4mL
   * Anesthesia protocol All surgery will be performed with standard general anesthesia. Induction will be achieved and general anesthesia maintained based on the following protocol

   (Doses vary based on patient specifics such as age, weight and comorbid disease): Lidocaine 50 - 100mg Fentanyl 50 - 100mcg Propofol 100 - 200 mg Rocuronium 50 - 100mg
   * Intraoperative:

   Sevoflurane 1 - 2% or desflurane 4 - 6% Fentanyl, hydromorphone, ketorolac and / or ketamine IV as needed on suspicion of pain.

   antibiotics were given intravenously 2g of cefazolin or 900mg of clindamycin.
   * Surgical procedure All surgery will be performed in beach chair position by a single shoulder and elbow fellowship trained surgeon. A standard deltopectoral approach will be used. A subscapularis peel-off will be used for all anatomic total shoulder arthroplasty cases and repaired back to the lesser tuberosity with transosseous sutures. For reverse shoulder arthroplasty cases, the subscapularis will be repaired if there is a reparable subscapularis tendon. Following the surgery, the shoulder will be immobilized in an abduction pillow-sling. A mixture of 1g of tranexamic acid and 30mL of normal saline will be poured into the wound for postoperative bleeding control purposes. Patients will follow the routine postoperative rehabilitation protocols. Patients will return to the shoulder and elbow clinic for routine clinical follow-up visits and x-ray exams following their surgery at 2 weeks, 6 weeks, 12 weeks, and 6 months, which is the standard of care. The study data collection will be completed at 2 week time point when the patient comes back for their first postoperative appointment.
   * Data collection: Following surgery, the patient's pain level will be recorded in a visual analog scale (VAS) at 4, 8, 12, 24 hours, once a day for the following 6 days, and at 14 days following surgery. Patient's daily opiate consumption during the first 7 days and the total cumulative amount of consumption up to 14 days following surgery will also be recorded, quantified and converted to morphine equivalents units (MEU) for standardization. Time to discharge from PACU as well as adverse opioid reactions will be reported (nausea, hypoxia/O2 requirement). The inpatient portion of the pain VAS and opiate consumption data will be obtained from the medical record while the post-discharge part of the data will be collected via a physical log given to patients upon discharge as well as an automated patient-reported outcome data collection system (PatientIQ®, Chicago, IL, USA). The research team will contact patients every other day following discharge to ensure proper documentation of pain VAS and opiate consumption by patients. Additionally, data regarding the time in the operating room, length of hospital stay, intraoperative complications (fracture, vascular injury, and anesthesia-related), acute postoperative complications (medical, nerve injury, dislocation, hematoma, and wound complications) will be collected. The average costs of LIA and interscalene regional block will be obtained through our billing department.

   Data analysis The pain score and opiate consumption data at each time point will be compared between the two groups using either unpaired t-test or Mann-Whitney U test depending on the data normality. The chronological changes in the pain score and opiate consumption in each patient will be analyzed using repeated measures ANOVA or Friedman test depending on the data normality. Categorical variables will be compared using chi-square test or Fisher's Exact test. The data will be analyzed by our biostatistics team within Department of Orthopaedic Surgery. The primary outcome of the study is the average pain VAS scores during the first 12 hours following surgery. The secondary outcome is the opioid consumption during the first 2 days following surgery. Non-inferiority of the local infiltration group compared to the interscalene block group in these two outcomes will be tested using a non-inferiority test.

   • Sample size calculation and power: The primary outcome of the study is the average pain VAS scores during the first 12 hours following surgery. Based on the recent research finding that a 1.4-point difference in pain VAS scores is a minimally clinically important difference (MCID) following shoulder arthroplasty, a priori sample size calculation was performed with a power of 0.8 and a standard deviation of 2.4 at an alpha of 0.05 to examine the study hypothesis that the average pain VAS score during the first 12 hours in the local infiltration analgesia group would not be significantly different than that of the interscalene block group (or the difference between the two groups would be less than 1.5 points). The result showed a minimum of 37 patients would be needed in each group (total number of patients =74).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or greater)
* Primary anatomic or reverse total shoulder arthroplasty secondary to osteoarthritis, cuff tear arthropathy, or massive irreparable rotator cuff tear

Exclusion Criteria:

* Narcotic dependent
* Previous ipsilateral open shoulder surgery
* Chronic pain syndromes (fibromyalgia)
* Contraindication to regional anesthesia
* Cervical radiculopathy
* Workers compensation insurance
* Mentally Disabled.
* Pregnant Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scale (VAS) | From 4 hours to 14 days postop
  Following surgery, the patient's pain level will be recorded in a visual analog scale (VAS) at 4 hours, 8 hours, 12 hours, 24 hours, 2 days and daily until 7 days, and then at 14 days.
Opiate consumption | From postop day 1 to 2 weeks
  The patient's daily opiate consumption during the first 7 days following surgery and the toal accumulated amount of opiate consumption by 2 weeks postop will also be recorded, quantified and converted to morphine equivalents units (MEU) for standardization

SECONDARY OUTCOMES:
Length of hospital stay | for postoperative 1 week
  Length of hospital stay
Postoperative complications | for postoperative 3 months
  Postoperative complications (medical, nerve injury, dislocation, hematoma, and wound complications)
Intraoperative complications | Intraoperative
  Intraoperative complications (fracture, vascular injury, and anesthesia-related),
Length of surgical procedure | Intraoperative
  Length of surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with other members of the research team.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared from actual study date until actual completion date
Access Criteria: * Treating relationship with a research team member listed on the IRB application.
  * Research team members will work directly with providers that have a treating (patient-provider) relationship

REFERENCES:
- [Result] Menendez ME, Lawler SM, Ring D, Jawa A. High pain intensity after total shoulder arthroplasty. J Shoulder Elbow Surg. 2018 Dec;27(12):2113-2119. doi: 10.1016/j.jse.2018.08.001. Epub 2018 Oct 12. PMID 30322752
- [Result] Bjornholdt KT, Jensen JM, Bendtsen TF, Soballe K, Nikolajsen L. Local infiltration analgesia versus continuous interscalene brachial plexus block for shoulder replacement pain: a randomized clinical trial. Eur J Orthop Surg Traumatol. 2015 Dec;25(8):1245-52. doi: 10.1007/s00590-015-1678-2. Epub 2015 Aug 15. PMID 26276164
- [Result] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Interscalene Block with and without Intraoperative Local Infiltration with Liposomal Bupivacaine in Shoulder Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2018 Aug 15;100(16):1373-1378. doi: 10.2106/JBJS.17.01416. PMID 30106818
- [Result] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Randomized Controlled Trial of Interscalene Block Compared with Injectable Liposomal Bupivacaine in Shoulder Arthroplasty. J Bone Joint Surg Am. 2017 Apr 5;99(7):550-556. doi: 10.2106/JBJS.16.00296. PMID 28375887
- [Result] Okoroha KR, Lynch JR, Keller RA, Korona J, Amato C, Rill B, Kolowich PA, Muh SJ. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: a prospective randomized trial. J Shoulder Elbow Surg. 2016 Nov;25(11):1742-1748. doi: 10.1016/j.jse.2016.05.007. Epub 2016 Jul 14. PMID 27422692
- [Result] Sabesan VJ, Shahriar R, Petersen-Fitts GR, Whaley JD, Bou-Akl T, Sweet M, Milia M. A prospective randomized controlled trial to identify the optimal postoperative pain management in shoulder arthroplasty: liposomal bupivacaine versus continuous interscalene catheter. J Shoulder Elbow Surg. 2017 Oct;26(10):1810-1817. doi: 10.1016/j.jse.2017.06.044. Epub 2017 Aug 24. PMID 28844420
- [Result] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Result] Sicard J, Klouche S, Conso C, Billot N, Auregan JC, Poulain S, Lespagnol F, Solignac N, Bauer T, Ferrand M, Hardy P. Local infiltration analgesia versus interscalene nerve block for postoperative pain control after shoulder arthroplasty: a prospective, randomized, comparative noninferiority study involving 99 patients. J Shoulder Elbow Surg. 2019 Feb;28(2):212-219. doi: 10.1016/j.jse.2018.09.026. Epub 2018 Dec 10. PMID 30545786
- [Result] Weller WJ, Azzam MG, Smith RA, Azar FM, Throckmorton TW. Liposomal Bupivacaine Mixture Has Similar Pain Relief and Significantly Fewer Complications at Less Cost Compared to Indwelling Interscalene Catheter in Total Shoulder Arthroplasty. J Arthroplasty. 2017 Nov;32(11):3557-3562. doi: 10.1016/j.arth.2017.03.017. Epub 2017 Mar 16. PMID 28390888
- [Result] Andersen LO, Kehlet H. Analgesic efficacy of local infiltration analgesia in hip and knee arthroplasty: a systematic review. Br J Anaesth. 2014 Sep;113(3):360-74. doi: 10.1093/bja/aeu155. Epub 2014 Jun 17. PMID 24939863
- [Result] Tashjian RZ, Hung M, Keener JD, Bowen RC, McAllister J, Chen W, Ebersole G, Granger EK, Chamberlain AM. Determining the minimal clinically important difference for the American Shoulder and Elbow Surgeons score, Simple Shoulder Test, and visual analog scale (VAS) measuring pain after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Jan;26(1):144-148. doi: 10.1016/j.jse.2016.06.007. Epub 2016 Aug 18. PMID 27545048